CLINICAL TRIAL: NCT02882139
Title: Multicenter Registry on Patients Affected by Electrical Storm
Brief Title: International Electrical Storm Registry
Acronym: ELECTRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Federico Guerra, Dr., Università Politecnica delle Marche
Other Study IDs: 2016-0364 OR
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Arrhythmias, Cardiac; Tachycardia, Ventricular; Ventricular Fibrillation; Defibrillators, Implantable
Keywords: Electrical storm
MeSH Terms: conditions — Arrhythmias, Cardiac; Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Electrical storm: Documentation of 3 or more episodes of sustained ventricular arrhythmia within 24h or documentation of sustained ventricular tachycardia lasted at least 12h

SUMMARY:
Organized ventricular arrhythmias (ventricular tachycardia (VT), torsades de pointes (TdP) and ventricular fibrillation (VF)) represent a major event in the clinical history of a patient and they can lead to hemodynamic instability and sudden cardiac death (SCD). Recurrences of ventricular arrhythmias and electrical instability have exponentially increased in the last decades and a new clinical entity called "electrical storm" (ES) has emerged as major morbidity and mortality factor. The ES is defined as a cluster of 3 or more sustained ventricular arrhythmias within 24 hours, or a sustained ventricular tachycardia lasting 12 hours or more and that does not respond to treatments.

Most of the patients presenting ES are already implanted with an ICD. This is due to 3 factors: first, patients with ICD implant are at higher risk to develop ventricular arrhythmias for the cardiac disease that led to the ICD implant. Second, the device records and treats also asymptomatic or poor symptomatic arrhythmic episodes that otherwise would not be detected. Third, and more important, the device gives the possibility to survive to an arrhythmic episode, making it possible for the patient to experience an ES. The incidence of ES is debated in different studies and ranges from 10 to 60% in patients with ICD for secondary prevention and from 4 to 7% in patients with ICD for primary prevention.

The aim of the ELECTRA registry is twofold:

1. To create an international registry on clinical features, optimal therapy, ablation strategy, prognosis and the effect of ICD programming on patients with ES.
2. To use the data derived from the registry for a prospective, observational study on mortality and rehospitalization rate in patients with ES.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ES (documentation of 3 or more episodes of sustained ventricular arrhythmia within 24h or documentation of sustained ventricular tachycardia lasted at least 12h).In order to fulfill this criterion, a patient with a previous episode of ES could also be enrolled during routine screening.
* Age ≥18
* Written informed consent

Exclusion Criteria:

* patient without ICD
* Confirmed or suspected use of drugs or narcotics with known direct pro-arrhythmic effect
* Inability to express an informed consent for the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be enrolled for a minimum of three years from the protocol approval. There is no pre-specified date for the end of enrollment, which will be decided by the study responsible according to the enrollment rate.
  A minimum of 500 patients will be included in the present registry. The exploratory nature intrinsic to the registry characteristics does not allow a sample size calculation by statistical means. However, the sample presented is based on the estimated enrolment rates of the participating centers during a 3-year enrolment period. Moreover, the sample size is large enough to postulate specific subgroup analyses.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Three years

SECONDARY OUTCOMES:
Hospitalization for all causes | Three years

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology and Arrhythmology Clinic, Marche Polytechnic University, University Hospital "Ospedali Riuniti", Ancona, Italy

REFERENCES:
- [Result] Guerra F, Palmisano P, Dell'Era G, Ziacchi M, Ammendola E, Bonelli P, Patani F, Cupido C, Devecchi C, Accogli M, Occhetta E, Santangelo L, Biffi M, Boriani G, Capucci A; Italian Association of Arrhythmology and Cardiac Pacing (AIAC). Implantable cardioverter-defibrillator programming and electrical storm: Results of the OBSERVational registry On long-term outcome of ICD patients (OBSERVO-ICD). Heart Rhythm. 2016 Oct;13(10):1987-92. doi: 10.1016/j.hrthm.2016.06.007. Epub 2016 Jun 9. PMID 27291511
- [Result] Guerra F, Flori M, Bonelli P, Patani F, Capucci A. Electrical storm and heart failure worsening in implantable cardiac defibrillator patients. Europace. 2015 Feb;17(2):247-54. doi: 10.1093/europace/euu298. Epub 2014 Oct 26. PMID 25345831
- [Result] Guerra F, Shkoza M, Scappini L, Flori M, Capucci A. Role of electrical storm as a mortality and morbidity risk factor and its clinical predictors: a meta-analysis. Europace. 2014 Mar;16(3):347-53. doi: 10.1093/europace/eut304. Epub 2013 Oct 4. PMID 24096960
- [Result] Guerra F, Palmisano P, Dell'Era G, Ziacchi M, Ammendola E, Pongetti G, Bonelli P, Patani F, Devecchi C, Accogli M, Occhetta E, Nigro G, Biffi M, Boriani G, Capucci A; Italian Association of Arrhythmology and Cardiac Pacing (AIAC). Cardiac resynchronization therapy and electrical storm: results of the OBSERVational registry on long-term outcome of ICD patients (OBSERVO-ICD). Europace. 2018 Jun 1;20(6):979-985. doi: 10.1093/europace/eux166. PMID 28595339
- [Result] Guerra F, Bonelli P, Flori M, Cipolletta L, Carbucicchio C, Izquierdo M, Kozluk E, Shivkumar K, Vaseghi M, Patani F, Cupido C, Pala S, Ruiz-Granell R, Ferrero A, Tondo C, Capucci A. Temporal Trends and Temperature-Related Incidence of Electrical Storm: The TEMPEST Study (Temperature-Related Incidence of Electrical Storm). Circ Arrhythm Electrophysiol. 2017 Mar;10(3):e004634. doi: 10.1161/CIRCEP.116.004634. PMID 28314850
- [Derived] Guerra F, Accogli M, Bonelli P, Carbucicchio C, Catto V, Cipolletta L, De Ferrari GM, Dell'Era G, Dusi V, Fabregat-Andres O, Flori M, Occhetta E, Palmisano P, Patani F, Proclemer A, Capucci A. IntErnationaL eLeCTRicAl storm registry (ELECTRA): Background, rationale, study design, and expected results. Contemp Clin Trials Commun. 2017 Jun 9;7:69-72. doi: 10.1016/j.conctc.2017.06.002. eCollection 2017 Sep. PMID 29696170

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT02882139/Prot_SAP_ICF_000.pdf